CLINICAL TRIAL: NCT02283931
Title: Assessement of Hemodynamic Changes Associated With Uterine Displacement Using Noninvasive Cardiac Output Monitoring and Transthoracic Echocardiography:
Brief Title: Cardiac Output Changes With Uterine Displacement
Acronym: LUDCO
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Awaiting New CoInvestigator with TTE Expertise
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Lawrence Ching Tsen, Associate Professor, Harvard Medical School, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014P002175
Record Dates: First submitted 2014-11-03; First posted 2014-11-05 (Estimated); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Obstetric Anesthesia, Cardiac Monitoring
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- One handed uterine displacement (Active Comparator): Uterine displacement using one hand
  Interventions: Device: TTE / NICOM
- two handed uterine displacement (Active Comparator): Uterine displacement using two hands
  Interventions: Device: TTE / NICOM
- 30 degrees uterine displacement (Active Comparator): Uterine displacement using a 30 degrees wedge
  Interventions: Device: TTE / NICOM

INTERVENTIONS:
Device: TTE / NICOM
  Other Names: Transthoracic Echocardiography / Noninvasive Cardiac Output Monitor

SUMMARY:
There is currently little information regarding the hemodynamic differences in uterine displacement techniques. Previous studies examining the hemodynamic effects of uterine displacement maneuvers have focused on incidence of hypotension and use of ephedrine.

Noninvasive cardiac output monitoring (NICOM) and transthoracic echocardiography (TTE) are becoming popular techniques in anesthesiology because they can provide noninvasive, valid, and precise hemodynamic data.There has been no study specifically examining the hemodynamic differences between the uterine displacement techniques using NICOM or TTE. While all three uterine displacement techniques are recommended, whether one technique may maximize maternal cardiac output is currently unknown.

DETAILED DESCRIPTION:
Aortocaval compression is a well-recognized physiologic concern in pregnancy. The gravid uterus can compress the inferior vena cava, impeding venous return and thereby reducing stroke volume and cardiac output.

The 2014 Society for Obstetric Anesthesia and Perinatology consensus statement on the management of cardiac arrest in pregnancy, and the 2010 American Heart Association guideline on maternal cardiac arrest recommend relieving aortocaval compression during chest compressions by performing uterine displacement There is currently little information regarding the hemodynamic differences amongst the recommended uterine displacement techniques. Previous studies examining the hemodynamic effects of uterine displacement maneuvers have focused on incidence of hypotension and use of ephedrine.

Noninvasive cardiac output monitoring (NICOM) and transthoracic echocardiography (TTE) are becoming popular techniques in anesthesiology because they can provide noninvasive, valid, and precise hemodynamic data.There has been no study specifically examining the hemodynamic differences between the uterine displacement techniques using NICOM or TTE. While all three uterine displacement techniques are recommended, whether one technique may maximize maternal cardiac output is currently unknown.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy ASA physical status I-II
2. Term parturient

Exclusion Criteria:

1. Woman in labor
2. Presence of maternal medical conditions affecting the cardiovascular system (including preeclampsia, gestational hypertension)
3. Fetal anomaly or intrauterine growth restriction (< 25th percentile)
4. Maternal renal or endocrine disease

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Cardiac Output | 10 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Bieniarz J, Yoshida T, Romero-Salinas G, Curuchet E, Caldeyro-Barcia R, Crottogini JJ. Aortocaval compression by the uterus in late human pregnancy. IV. Circulatory homeostasis by preferential perfusion of the placenta. Am J Obstet Gynecol. 1969 Jan 1;103(1):19-31. doi: 10.1016/s0002-9378(16)34335-6. No abstract available. PMID 5761773
- [Result] Bamber JH, Dresner M. Aortocaval compression in pregnancy: the effect of changing the degree and direction of lateral tilt on maternal cardiac output. Anesth Analg. 2003 Jul;97(1):256-8, table of contents. doi: 10.1213/01.ane.0000067400.79654.30. PMID 12818977
- [Result] Lewis JF, Kuo LC, Nelson JG, Limacher MC, Quinones MA. Pulsed Doppler echocardiographic determination of stroke volume and cardiac output: clinical validation of two new methods using the apical window. Circulation. 1984 Sep;70(3):425-31. doi: 10.1161/01.cir.70.3.425. PMID 6744546
- [Result] Dennis A, Stenson A. The use of transthoracic echocardiography in postpartum hypotension. Anesth Analg. 2012 Nov;115(5):1033-7. doi: 10.1213/ANE.0b013e31826cde5f. Epub 2012 Oct 9. No abstract available. PMID 23051881